CLINICAL TRIAL: NCT06798935
Title: Feasibility and Safety of Additional Injection of Autologous Platelet-rich Stroma to Surgical Treatment of Rectovaginal Fistulas
Acronym: PRS-RVF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: IJsselland ziekenhuis (Unknown)
Responsible Party: Principal Investigator, Anne S. Nieuwstraten, BSc, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEC-2019-0038
Record Dates: First submitted 2025-01-18; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Rectovaginal Fistula; Anovaginal Fistula
Keywords: rectovaginal fistula; anovaginal fistula; platelet-rich stroma; stromal vascular fraction; platelet-rich plasma; autologous; cell therapy
MeSH Terms: conditions — Rectovaginal Fistula

STUDY DESIGN:
Intervention Model Description: Prospective cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Additional PRS-injection (Experimental): Patients suffering from rectovaginal fistula's underwent rectovaginal fistula surgery with an additional injection of autologous PRS
  Interventions: Procedure: autologous platelet-rich stroma

INTERVENTIONS:
Procedure: autologous platelet-rich stroma — Autologous platelet-rich stroma, which is the combined product of stromal vascular fraction and platelet-rich plasma

SUMMARY:
Is the addition of platelet-rich stroma (PRS) injection, a form of autologous call therapy, to surgical treatment for rectovaginal fistula feasible and safe? The primary endpoints of this study are feasibility and safety until 12 months after surgery. Secondary endpoints include rates of clinical and radiological closure, recurrence rates after clinical or radiological closure and unplanned re-interventions within 12-month post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients presenting with significant symptoms of a rectovaginal fistula (RVF)
* RVF confirmed on imaging or with a high suspicion based on imaging findings (magnetic resonance imaging [MRI] and/or endoanal ultrasound [EUS])

Exclusion Criteria:

* Patients with active proctitis
* Patients with the presence of associated (not properly drained)) pelvic abscess
* Patients with immune suppressed status
* Patients with hematological disorders
* Patients with any oncological event in the five years prior to study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-01-11 (Actual); Primary Completion 2024-09-04 (Actual); Study Completion 2024-09-04 (Actual)

PRIMARY OUTCOMES:
Number of patietns with feasible PRS injection | 1 day (day of surgery)
  Feasibility was assessed by the ability to successfully obtain SVF and PRP and to inject the combined product (i.e. PRS) during the procedure.

SECONDARY OUTCOMES:
Number of patients with safe PRS injection | 30 days postoperatively
  Safety was assessed by documenting the number of (serious) adverse events related to PRS injection within 30 days postoperatively. In addition, we report on number of serious fistula-related emergency room (ER) visits and number of readmissions within 30 days postoperatively.
Number of patients with clinical closure | 12 months
  closure of the vaginal fistula opening without complaints of discharge at physical examination
Number of re-interventions | 12 months
  ) the need for unplanned re-interventions due to residual clinical and/or radiological fistulizing disease or recurrent disease
Number of patients with radiological healing | 12 months
  radiological healing or radiological improvement, based on available MRI reports
Number of patients with recurrence | 12 months
  the reopening of the vaginal fistula opening after clinical closure and/or radiological healing

CONTACTS AND LOCATIONS:
Overall Officials: Oddeke van Ruler, GI- surgeon, MD, PhD, Principal Investigator — IJsselland Hospital
Locations (1):
- Ijsselland Hospital, Capelle aan den IJssel, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Deijl W, Arkenbosch J, van Ruler O, van der Woude CJ, Stevens HPJD, de Graaf E, Schouten R. Autologous Platelet-Rich Stroma in Complex Perianal Fistulas. Dis Colon Rectum. 2020 Jun;63(6):860-861. doi: 10.1097/DCR.0000000000001546. No abstract available. PMID 32384409
- [Background] Schouten WR, Arkenbosch JHC, van der Woude CJ, de Vries AC, Stevens HP, Fuhler GM, Dwarkasing RS, van Ruler O, de Graaf EJR. Efficacy and safety of autologous adipose-derived stromal vascular fraction enriched with platelet-rich plasma in flap repair of transsphincteric cryptoglandular fistulas. Tech Coloproctol. 2021 Dec;25(12):1301-1309. doi: 10.1007/s10151-021-02524-6. Epub 2021 Oct 4. PMID 34606026
- [Background] Arkenbosch JHC, van Ruler O, Dwarkasing RS, Fuhler GM, Schouten WR, van Oud-Alblas MB, de Graaf EJR, de Vries AC, van der Woude CJ. Stromal vascular fraction with platelet-rich plasma injection during surgery is feasible and safe in treatment-refractory perianal fistulising Crohn's disease: A pilot study. Aliment Pharmacol Ther. 2023 Apr;57(7):783-791. doi: 10.1111/apt.17347. Epub 2022 Dec 26. PMID 36571818